CLINICAL TRIAL: NCT03833492
Title: Efficacy and Safety of Underwater vs. Conventional Endoscopic Mucosal Resection for the Treatment of Diminutive Non-pedunculated Colorectal Polyps：A Multicenter Randomized Clinical Trial
Brief Title: UEMR vs. CEMR for Diminutive Non-pedunculated Colorectal Polyps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ningbo No. 1 Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UEMR-1.0
Record Dates: First submitted 2019-02-04; First posted 2019-02-07 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Colonic Polyps
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Underwater EMR (Experimental): The patients who are randomized to the " Underwater EMR" arm polypectomy with water will be performed under full water emersion without the use of submucosal injection.
  Interventions: Behavioral: Underwater EMR
- Traditional EMR (No Intervention): The patients who are randomized to the " Traditional EMR" arm polypectomy will be performed with selective saline injection to the layer of tissue underneath the polyp in order to create a "safety cushion" for resection.

INTERVENTIONS:
Behavioral: Underwater EMR — Polypectomy is performed under full water emersion without the use of submucosal injection.
  Arms: Underwater EMR

SUMMARY:
This clinical trial is being conducted to compare the efficacy and safety of two standard methods of polypectomy，Conventional Endoscopic Mucosal Resection（EMR）and Underwater Endoscopic Mucosal Resection（UEMR），for small colorectal polyps.

ELIGIBILITY:
Inclusion Criteria:

Patients age between 18-75 years old with non-pedunculated colonic polyps (measuring between 4 and 9mm), who willing to participate in this study.

Exclusion Criteria:

1. pregnancy,
2. inflammatory bowel disease,
3. familial polyposis
4. the use of anticoagulant therapy or antiplatelet therapy
5. the absence of informed patient consent.
6. Polyps showing signs of deep submucosal invasion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-12 (Actual)

PRIMARY OUTCOMES:
complete resection rate | 7 days
  complete resection rate is defined as a complete en bloc resection of a lesion with tumor-free lateral and vertical margins.
En bloc resection rate | immediately
  En bloc resection rate was defined as the entire lesion could be removed in 1 piece instead of piecemeal resection.

SECONDARY OUTCOMES:
Adverse event rate | 14 days
  Including bleeding and perforation , etc.
Procedure time | 24 hours
  Time to execute the program

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Department of Gastroenterology, Haishu No.2 Hospital, Ningbo, China, Ningbo, Zhejiang
  - Department of Gastroenterology, Ninghai No.2 Hospital, Ningbo, China, Ningbo, Zhejiang
  - Ningbo first hospital, Ningbo, Zhejiang

REFERENCES:
- [Derived] Zhang Z, Xia Y, Cui H, Yuan X, Wang C, Xie J, Tong Y, Wang W, Xu L. Underwater versus conventional endoscopic mucosal resection for small size non-pedunculated colorectal polyps: a randomized controlled trial : (UEMR vs. CEMR for small size non-pedunculated colorectal polyps). BMC Gastroenterol. 2020 Sep 23;20(1):311. doi: 10.1186/s12876-020-01457-y. PMID 32967616